CLINICAL TRIAL: NCT06805708
Title: Educational Intervention for Sleep Hygiene Nursing in Adolescents: Translation to the School Nurse
Brief Title: Educational Intervention for Sleep Hygiene Nursing in Adolescents
Acronym: ENISHA-ST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5481
Record Dates: First submitted 2025-01-17; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: School-based Intervention; Sleep
Keywords: School setting; Sleep pattern; Physical activity; Nursing; Health Promotion; Prevention and monitoring; Participatory action research
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participatory Action Research (PAR) focusing on cognitive-behavioural counselling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep hygiene training programme (Experimental): A programme focusing on cognitive-behavioural counselling. The programme will be delivered in 12 sessions of 30 minutes each (intensive phase: 1 session per week for 3 weeks; maintenance phase: 1 session every 2 weeks). The discussion topics will be the management of sleep hygiene in schoolchildren, families and teachers, and educational elements.
  Interventions: Behavioral: Sleep hygiene training programme

INTERVENTIONS:
Behavioral: Sleep hygiene training programme — A programme focusing on cognitive-behavioural counselling. The programme will be delivered in 12 sessions of 30 minutes each (intensive phase: 1 session per week for 3 weeks; maintenance phase: 1 session every 2 weeks). After each meeting, the research group members will provide a short-written report reflecting the main discussion topics, the degree of participation, and the group's position in the participatory action research cycle. The discussion topics will be:
  1. Management of sleep hygiene in schoolchildren, families and teachers:
     * Surveys (quantitative approach)
     * Focus groups (qualitative approach)
     * The study will identify the health assets
  2. Educational elements

SUMMARY:
There is an urgent need to influence the knowledge and beliefs associated with sleep (TV viewing, use of electronic devices, sedentary activity...) of school children through holistic interventions involving students, parents, teachers and other professionals in the education sector that can positively influence education. The project's main objective is to determine the acceptability and effectiveness of a school intervention consisting of counselling by family and community nurses. The methodological approach is Participatory Action Research (PAR), developed in three phases: exploratory, intervention, and evaluation. In the exploratory phase, which corresponds to a research study with a qualitative (focus groups and content analysis) and quantitative (questionnaires) approach, the study subjects will be students in the second year of secondary education in five schools in southern Spain (city and province), as well as parents and teachers. Sampling will be probabilistic. Following the action research cycle, the results of the exploration phase will be shared with all participants and will be considered for the intervention phase. This phase will aim to conceptualise/implement a sleep hygiene programme. It will take into account key aspects such as (i) health education, (ii) sleep hygiene, (iii) breathing control to facilitate sleep, (iv) sleep restriction, and (v) stimulus control. The programme will be implemented during 12 sessions of 30 minutes (intensive phase: 1 session/week for 3 weeks; maintenance phase: 1 session every 2 weeks) and will focus on cognitive-behavioural counselling. The intervention will be applied to the referred students from the participating schools. For this phase, the data analysis will be quantitative (pre-post intervention). The evaluation phase will occur 6 and 12 months after the intervention, with the same methodological approach as in the exploratory phase (quantitative and qualitative).

ELIGIBILITY:
Inclusion Criteria:

* All schoolchildren aged between 13-16 years who provide signed consent and participation by their parents/legal guardian.
* Schoolchildren taking medication that interferes with the sleep/wakefulness pattern or presenting pathologies that alter the sleep pattern (respiratory, digestive...) will also be considered.
* Family members of schoolchildren and teaching staff who agree to participate in the study will be included.

Exclusion Criteria:

* Failure to sign the informed consent and participation form

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Sleep hygiene (Adolescent Sleep Hygiene Scale) | From enrollment to through study completion, an average of 1 academic year
  The ASHS is a 32-item self-report measure used to assess adolescent sleep hygiene (LeBourgeois et al., 2005). The ASHS includes four qualitative items to ascertain usual bedtime and wake time on weekdays and weekends and 28 quantitative items that are used to calculate nine subscale scores: physiological (5 items), cognitive (6 items), emotional (3 items), sleep environment (4 items), daytime sleep (1 item), substances (2 items), sleep stability (4 items), bedtime routine (1 item) and bed sharing (2 items). Response choices are on a 6-point ordinal scale: 1 = Never (0%); 2 = Once in a while (20%); 3 = sometimes (40%); 4 = quite often (60%); 5 = frequently, if not always (80%); 6 = always (100%). Scoring: Each subscale score is calculated by taking the average of the items comprising that subscale.
Sleep quality (Pittsburgh Sleep Quality Index) | From enrollment to through study completion, an average of 1 academic year
  The questionnaire consists of a combination of Likert-type and open-ended questions. Respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Sleep duration (sleep diaries) | From enrollment to through study completion, an average of 1 academic year
  Sleep diary includes entries for bedtimes, wake-up times, the number and duration of awakenings during the night, overall sleep duration, perceived quality of sleep, and daily activities that might affect sleep, such as caffeine or alcohol intake, exercise, and naps.

SECONDARY OUTCOMES:
Socio-cognitive determinants | From enrollment to through study completion, an average of 1 academic year
  Knowledge, attitude, subjective norm, perceived behavioural control and intention. The Sleep Knowledge Questionnaire (SKQ) scores from 0 to 20, where higher points reflect sleep knowledge. The Sleep Attitudes Questionnaire uses a 5-point Likert scale (10 to 50 points), with higher scores indicating favourable attitudes toward sleep. The Subjective Norm Scale typically has a 7-point scale (7 to 49 points) reflecting perceived social pressure. The Self-Efficacy for Sleep Scale is scored on a 10-point scale (10 to 100 points), where higher scores show more confidence in sleep management. Finally, the Sleep Intention Scale employs a 5-point scale (5 to 25 points), with higher scores signifying greater intentions to adopt positive sleep behaviours.
Sociodemographic, family, and lifestyle and habits | From enrollment to through study completion, an average of 1 academic year
  The research team will create a questionnaire to capture relevant variables. Participants will report sociodemographic factors like age (age ranges), sex (male, female, other), and perceived social class (lower, middle, upper). Family variables will include cohabitation status (living alone, with family, with friends) and the number of family members (1, 2-3, 4 or more). Lifestyle questions will cover physical activity levels (sedentary, moderate, active), eating habits (balanced, unhealthy, irregular), hygiene practices (daily, weekly), and substance use (none, occasional, regular tobacco, alcohol, or other drugs).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Maimónides de Investigación Biomedica de Cordoba, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol